CLINICAL TRIAL: NCT06149455
Title: A Randomized Controlled Trial of Preoperative Prophylactic Antibiotics for Ureteroscopy in Moderate to High Infectious Risk Population
Brief Title: Preoperative Prophylactic Antibiotic Duration in Moderate to High Risk Ureteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-37824
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Infections, Urinary Tract; Nephrolithiasis
MeSH Terms: conditions — Urinary Tract Infections; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short duration of preoperative antibiotics (2 days) (Experimental)
  Interventions: Other: Duration of antibiotics
- Long duration of preoperative antibiotics (7 days) (Active Comparator)
  Interventions: Other: Duration of antibiotics

INTERVENTIONS:
Other: Duration of antibiotics — Patients will be randomized to a short (2 days) or long (7 days) of pre-operative antibiotics, the choice of agent will be dependent upon bacterial sensitivities if available which is standard of care.

SUMMARY:
The goal of this non-inferiority randomized controlled trial: is to test the hypothesis that the that there is no additional benefit from a longer course (7 days) versus a shorter course (2 days) of pre-operative antibiotics in patients with moderate to high risk of infection undergoing ureteroscopy. The main questions it aims to answer are:

1. Determine the safety and efficacy of a short course (2 days) as compared to a long course (7 days)
2. Identify secondary predictors of post-operative infectious complications

DETAILED DESCRIPTION:
Post-operative infectious complications including urinary tract infection (UTI), systemic inflammatory response syndrome (SIRS), and sepsis are uncommon but potentially devastating complications after ureteroscopy. The clinical guidance from the American Urologic Association (AUA) and the European Association of Urology (EAU) is to provide treatment for symptomatic urinary tract infections however the management for asymptomatic patients with positive cultures or those patients who are otherwise at high risk of urinary tract colonization is unclear. As a result, there is significant practice variation in pre-operative prophylactic antibiotic prescription, even amongst fellowship trained endourologists, with some providers prescribing over ten days of pre-operative antibiotics while others offer none. This is a critical gap in our understanding of pre-operative prophylactic antibiotic utilization in a population of patients not only at higher risk of harboring multi-drug resistant (MDR) organisms but are also more susceptible to deleterious outcomes due to their frailty. Recent randomized trials have demonstrated that short courses of pre-operative antibiotics are no less protective than long courses in patients undergoing percutaneous nephrolithotomy (PCNL) for stone removal. Ureteroscopy is the most commonly performed stone surgery worldwide. Establishing an evidence-based approach for antibiotic prophylaxis in the ureteroscopic surgical patient population will be impactful for a large number of patients. The goal of this study is to implement a well-designed randomized clinical trial to establish the standardized antibiotic protocol necessary to minimize unnecessary antibiotic use which may otherwise lead to adverse reactions and proliferation of multi-drug resistant organisms.

ELIGIBILITY:
Inclusion Criteria:

* age (greater than or equal to 18 years)
* indwelling ureteral stent in place
* nephrostomy tube in place
* indwelling foley catheter, suprapubic catheter or clean intermittent catheterization
* asymptomatic bacteriuria
* bowel interposition (such as ileal conduit, neobladder)
* immunosuppression (such as for transplant recipients, active chemotherapy use)

Exclusion Criteria:

* pregnancy
* active infection
* received antibiotics within 7 days preceding surgery that were not prescribed for the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
infectious complication rate | 30 days after surgery
  any occurrence of urinary tract infection, pyelonephritis, systemic inflammatory response syndrome or sepsis

SECONDARY OUTCOMES:
Non-infectious complications including readmission | 30 days after surgery
  Any other complications after the surgical procedure such as pain, readmission, urinary retention, etc
Adverse reaction to antibiotic regimen | 2-7 days prior to surgery (depending on which arm the patient was randomized to)
  Any adverse reaction to antibiotic regimen
Identification of secondary markers of post-operative sepsis | Obtained during the peri-operative period
  Markers of infection will be drawn preoperatively including erythrocyte sedimentation rate, c-reactive protein test, intra-operative renal pelvis pressure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
We have no plans to make individual participant data available to other researchers.